CLINICAL TRIAL: NCT04311112
Title: Safety and Efficacy of Zuretinol Acetate Oral Solution in Subjects With Inherited Retinal Disease Caused by Mutations in Retinal Pigment Epithelium Protein 65 or Lecithin:Retinol Acyltransferase
Brief Title: Safety and Efficacy of Zuretinol Acetate in Subjects With Inherited Retinal Disease
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The asset was transferred to another company
Sponsor: Retinagenix Holdings (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RG201
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2020-10

CONDITIONS: Retinal Disorder
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ZA placebo (Placebo Comparator)
  Interventions: Drug: Placebos
- ZA low dose (Active Comparator)
  Interventions: Drug: ZA Low dose
- ZA high dose (Active Comparator)
  Interventions: Drug: ZA high dose

INTERVENTIONS:
Drug: Placebos — Placebo
  Arms: ZA placebo
Drug: ZA Low dose — ZA low dose
  Arms: ZA low dose
Drug: ZA high dose — ZA high dose
  Arms: ZA high dose

SUMMARY:
To evaluate the efficacy of ZA oral solution in subjects with IRD caused by biallelic recessive RPE65 or LRAT gene mutations and phenotypically diagnosed as Leber's Congenital Amaurosis (LCA) or Retinitis Pigmentosa (RP).

ELIGIBILITY:
Inclusion Criteria:

1. Have read, understood and signed the informed consent form (ICF).
2. Be aged 6 years or older.
3. Have a diagnosis of IRD phenotypically diagnosed as LCA or RP by an ocular geneticist or ophthalmologist and caused by pathologic biallelic autosomal recessive mutation in RPE65 or LRAT as determined by a fully accredited certified central genotyping laboratory.
4. Be naïve to gene therapy, surgical implantation of prosthetic retinal chips, or subretinal injections.
5. If previously administered ZA , have at least > 3 years since last administration of ZA.
6. Pregnancy testing and contraception before study treatment: Women of childbearing potential must not be pregnant or lactating.

Exclusion Criteria:

1. Have a presence of concurrent ocular disease that in the opinion of the Investigator would put the subject at greater risk during the study or significantly affect study results.
2. Have had ocular surgery within 3 months of Screening, including cataract or laser procedures.
3. Have taken any prescription or investigational oral retinoid medication (e.g., isotretinoin or acitretin) within 6 months of Screening; subjects who did not tolerate their previous oral retinoid medication will be excluded regardless of the time of last exposure.
4. Have taken any supplements containing ≥ 10,000 IU vitamin A within 60 days of Screening.
5. Have taken any medication that affects bone metabolism within 6 months of Screening.
6. Have circulating 25-hydroxy vitamin D < 20 ng/mL.
7. Use of medications that may interact with a retinoid, including tetracycline, ketoconazole and methotrexate within 60 days of Screening.
8. Use of intraocular or periocular corticosteroids within 90 days of Screening; use of corticosteroid implants within 3 years of Screening; use of systemic corticosteroids unless these are at a steady low dose with low dose level in effect prior to or at Screening; or use of intraocular or periocular anti-vascular endothelial growth factor agents within 2 months of Screening.
9. Have a known and documented allergy to soy.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in functional vision at Week 12 using a visual navigation course at different ambient illumination levels | week 12
  The primary efficacy endpoint (PEE) will be a measure of functional vision assessed at Week 12 employing mobility testing (Ora Inc, Andover, MA) via their Visual Navigation Challenge (VNC) course. The VNC measures functional vision by evaluating the subject's ability to navigate a maze accurately and successfully at different levels of ambient illumination. The PEE is a comparison between groups in their mean change from randomization to week 12, that is, the difference in VNC score from baseline performance to week 12 performance. Performance on the VNC is assessed using each eye individually and both eyes together at 1 or more levels of illumination that range from 0.35 lux to 500 lux. A subject's VNC score is the lowest level of luminance at which the subject can navigate and correctly pass through the maze.

CONTACTS AND LOCATIONS:
Locations (1):
- NY NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No